CLINICAL TRIAL: NCT05378568
Title: Implementation and Evaluation of the Selection Scheme of Peripheral Venous Infusion Devices for Hospitalized Children: a Stepped Wedge Cluster Randomized Trial
Brief Title: Implementation and Evaluation of the Selection Scheme of Peripheral Venous Infusion Devices for Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FNF202112
Record Dates: First submitted 2022-02-23; First posted 2022-05-18 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Children,Hospitalized; Vascular Access Devices
Keywords: pediatric; implementation study; peripheral venous access devices; selection; effect evaluation; appropriateness; randomised trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the selection scheme of peripheral venous access devices (Experimental): To implement the selection scheme of peripheral venous access devices, based on the Clinical Practice Guideline on Infusion Therapy in Children. Then observe the appropriateness of peripheral venous access devices selection.
  Interventions: Other: the selection scheme of peripheral venous access devices
- the existing nursing routine (Active Comparator): Follow the existing nursing routine of intravenous infusion and the selection of peripheral venous access devices.
  Interventions: Other: the existing nursing routine

INTERVENTIONS:
Other: the selection scheme of peripheral venous access devices — Based on the "Facilitator Toolkit" of the promoting action on research implementation in health services integrated framework(i-PARIHS), the implementation plan of peripheral intravenous infusion device selection in hospitalized children was formulated and applied, so as to change the practice behavior of nurses in the intervention group. The specific process mainly includes: tailoring evidence; baseline review; situational analysis; promotion and implementation strategy like lectures, group discussions, operation demonstrations, and scenario simulations.
  Arms: the selection scheme of peripheral venous access devices
Other: the existing nursing routine — To choose infusion device according to nurse's working experience. First, nurse placed a peripheral intravenous catheter. The patients and family decide whether to place the central intravenous infusion device according to the recommendation of the medical staff.
  Arms: the existing nursing routine

SUMMARY:
This study is a stepped wedge cluster randomized trial design. The object is to evaluate the influence on patient outcomes, medical staff's evidence-based practice behavior and hospital context after implementation of the selection scheme of venous access devices comes from" Evidence-based guidelines for clinical practice of intravenous infusion therapy in children". This study sought to compare the appropriateness of peripheral venous access device selection, to compare the incidence of infiltration and extravasation and the cost of venous infusion consumables before and after the implementation of the scheme.

DETAILED DESCRIPTION:
This study aimed to improve the standardization and suitability of device use and reduce complications associated with intravenous fluids by implementing best practice evidence for intravenous fluid device selection in children. In 2021, the Chinese Journal of Evidence-Based Pediatrics released the " Evidence-based guidelines for clinical practice of intravenous infusion therapy in children". The researchers used the evidence in this guideline as a standard to understand the current status of clinical intravenous infusion device selection and the gap between the current situation and the evidence. The evidence tailor, baseline review, develop implementation plan, conduct implementation research. A stepped wedge cluster randomized trial divided into 5 steps, 10 clusters(units), and the step size was one month. Each included ward of a tertiary first-class pediatric hospital was regarded as a group, and each step was included into randomized two groups, and the observation was maintained for one month until all units were included in the intervention in the fifth month, with a total of 6 research periods. Given the practicality of the study design, limited additional inclusion and exclusion criteria will be added.

ELIGIBILITY:
Inclusion Criteria for nurses:

* Nurses have been working in the siting more than 1 year
* Nurses who can independently perform nursing operations (complete the contents related to intravenous infusion in the standardized training of hospital and pass the examination)

Inclusion Criteria for patients:

* Patients receiving intravenous infusion
* Hospitalized patients aged 28 days to 18 years

Exclusion Criteria for nurses:

* Nurses who has not obtained the practicing qualification certificate
* Nurses refused to participate in the study

Exclusion Criteria for patients:

* The indwelling time is less than 24h
* Patients who were put into intravenous catheter at admission and did not receive new catheter during hospitalization
* Patients with only one stat(st) order for intravenous infusion during hospitalization
* Patients refused to participate in the study

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4652 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Error rate in peripheral intravenous infusion device selection | 6 months
  The selection is made according to the recommendation of the guidelines. Those who conform to the recommendation are correct, those who do not conform are wrong. Calculation method: the error rate = (the number of cases with wrong peripheral intravenous infusion device selection)/(the total number of cases using peripheral intravenous infusion device)* 100%.

SECONDARY OUTCOMES:
The knowledge level of nurses' intravenous infusion device selection | 6 months
  The questionnaire has a total of 50 questions, 24 choice questions, 12 judgment questions, and 14 fill-in-the-blank questions, each with 2 points, and the total score is 100 points. Before and after the implementation of the program, the evaluation will be conducted, a score of less than 60 is considered a failure, and a score of more than 80 is considered excellent.
Compliance of evidence-based practice behavior of nurses | 6 months
  compliance of each review indicator = (the number of correct implementation of this indicator by nurses)/(the total number of reviews of this indicator) *100%
Incidence of infiltration and/or extravasation | 6 months
  The bedside nurses document the number of incidents of peripheral venous infiltration and extravasation using "Pediatric Peripheral Venous Infiltration Scale". The incidence of infiltration and/or extravasation = (case numbers of infiltration and/or extravasation)/(Catheter Days per Month)×1000‰.
The cost of intravenous infusion consumables | 6 months
  including intravenous infusion devices (including the total number of catheters consumed by successful catheter placement and failed puncture), dress, central venous maintenance kits, infusion connectors, and tees.
Implementation process evaluation based on "Reach*Efficacy(RE)-Adoption, Implementation, and Maintenance(AIM)" framework | 6 months
  including Reach, Efficacy, Adoption, Implementation, and Maintenance. Reach refers to the participation rate of training courses; Efficacy refers to the change of knowledge level and compliance of evidence-based practice behavior of nurses in the intervention group; Adoption refers to the proportion of evidence actually adopted by nurses in the intervention group and the changes of context; Implementation refers to the completion rate of each training plan in the implementation strategy；Maintenance refers to evaluating the maintenance of the selection scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No